CLINICAL TRIAL: NCT02155894
Title: Tight Control of Disease Activity Among Patients With Rheumatoid Arthritis Based on a Systematic Telemedicine Treatment Strategy
Brief Title: Tight Control of Disease Activity Among Patients With RA Based on a Systematic Telemedicine Treatment Strategy
Acronym: TeRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: TeRA_15-05-14
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis, treat to target, telemedicine
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Telemedicine; Nurses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Disease control, Telemedicine, doctor (Experimental): Using an online platform for self assessment and with the Flare instrument as decision support, the patients are contacted over the telephone by a doctor at week 13, 26, 39.
  Interventions: Behavioral: Disease control, Telemedicine, doctor
- Disease control, Telemedicine, nurse (Experimental): Using an online platform for self assessment and with the Flare instrument as decision support, the patients are contacted over the telephone by a nurse at week 13, 26, 39.
  Interventions: Behavioral: Disease control, Telemedicine, nurse
- Usual care (No Intervention): Usual care: control of disease activity with consultations in the outpatient clinic.

INTERVENTIONS:
Behavioral: Disease control, Telemedicine, doctor — Control of disease activity by a telemedicine consultation carried out by a doctor.
  The telemedicine consultation will be based on a telephone consultation, following a predefined consultation checklist.
  Patients who have expressed a desire to complete questionnaires in webform, will receive a letter a week before the consultation to remind them that they must assess their disease activity through the software interphase, within the next couple of days. Patients, who have expressed a wish to fill in questionnaires in paperform, will receive the questionnaire a week before the consultation.
  During telephone consultation, updated clinical test results will be available through the electronic medical system.
  Arms: Disease control, Telemedicine, doctor
Behavioral: Disease control, Telemedicine, nurse — Control of disease activity by a telemedicine consultation carried out by a nurse.
  The telemedicine consultation will be based on a telephone consultation, following a predefined consultation checklist.
  Patients who have expressed a desire to complete questionnaires in webform, will receive a letter a week before the consultation to remind them that they must assess their disease activity through the software interphase, within the next couple of days. Patients, who have expressed a wish to fill in questionnaires in paperform, will receive the questionnaire a week before the consultation.
  During telephone consultation, updated clinical test results will be available through the electronic medical system.
  Arms: Disease control, Telemedicine, nurse

SUMMARY:
The study aims to investigate the effect a systematic telemedicine intervention, based on the tigth control principals, as a platform for disease monitoring among patients with rheumatoid arthritis.

It is hypothesized that:

* A systematic telemedicine intervention targeted to tight control of disease activity among patients with RA will be equally effective as usual care (outpatient consultation by a rheumatologist).
* There will be no difference in the effect whether this telemedicine consultation is carried out by a rheumatologist or a rheumatology nurse.
* Patient satisfaction and the patient's general perception of involvement in their treatment will be increased for patients who receive the telemedicine intervention.
* All the effects will apply both in the short term (< 6 months) and in the long term (> 1 year).

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic disease affecting 0.5-1.0 % of the Danish population. Due to an expected growing population and a higher proportion of elderly the prevalence is likely to increase in the years to come.

Untreated RA will lead to joint destruction disabling the patients, but in recent years both treatment and treatment strategies have been markedly improved. According to international guidelines early start of medical treatment, quick escalation of doses, and adjustment of the dose throughout the whole disease course when there are signs of disease activity, are considered important elements in the RA treatment strategy. Consequently, the success of this strategy implies the possibility of regular routine testing of all RA patients, which could become a challenge to the health care system causing substandard treatment to RA patients in the future. This calls for reorganization of the routine care of RA, i.e. in form of a telemedicine intervention.

Telemedicine is considered to be the use of communication and information technologies to deliver clinical care where the individuals involved are not at the same location. No studies have yet investigated the effect of monitoring disease activity through a standardized telemedicine treatment strategy in patients with RA, and most of the evidence is derived from studies within chronic heart disease, chronic obstructive lung disease, asthma, diabetes and hypertension. This evidence indicates, however, that telemedicine interventions seem to be effective, time saving and associated with a high degree of patient satisfaction.

RA disease activity is measured using a composite score that includes both objective and subjective outcome parameters to measure present as well as past disease activity. These scores include: tender and swollen joint count together with the patient's global assessment, report of physical functioning, the measurement of an acute-phase reactant and serial radiographic assessment. The most commonly used instruments for measuring RA disease activity in daily clinical practice is the European League Against Rheumatism (EULAR) criteria, the Disease Activity Score 28 (DAS28).

However, in a telemedicine intervention there is no direct physical contact between the patient and the health professionals, making traditional disease activity measures unfit for use, as they imply an assessment of tender and swollen joints carried out by a health professional. It has been suggested to let the patients examine their joints. Still, it has been shown that patients tend to overestimate the presence of swollen joints which impairs the identification of synovitis - and thereby disease activity and flare. Hence, telemedicine disease activity monitoring in RA may be best supported by validated measures based on other kinds of patient self-assessment, i.e. the newly developed "Flare" instrument.

According to international recommendations from the European League Against Rheumatism (EULAR) patients should have access to nurse-led telephone services to enhance continuity of care and to provide ongoing support, but it still remains unclarified which of the occupational groups, doctors or nurses, is to carry out the routine telemedicine disease monitoring.

The trend in RA treatment is towards patients taking a more active role in the treatment, and telemedicine could be a very workable solution. However, before decision is made of transforming tight control of disease activity among patients with RA into a telemedicine intervention the effectiveness of such intervention, both when executed by doctors and nurses, need to be investigated.

The objectives of this study are:

1. To test the effectiveness of a customized telemedicine intervention targeted to tight control of disease activity among patients with RA, compared with usual outpatient care in a pragmatic randomized controlled trail.
2. To test if the effect differs depending on whether the telemedicine consultation is carried out by a rheumatologist or by a rheumatology nurse.
3. To examine the patients perspective towards telemedicine tight control of disease activity in RA, and assess patient satisfaction and acceptability towards the intervention.

Power calculation

A decrease in DAS28 on 1.2 is regarded as a significant clinically improvement. A change in DAS28 on 0.6 is regarded as non-response . Thus, a change in the DAS28 score >0.6 will be used as the cut-point for a change in the condition. The standard deviation in DAS28 is presumed to be 1.5. Hence, in order to detect a 1-sided statistically significant change between the three groups, with a statistical power on 80% (beta=0.20), a sample size of at least 98 patients in each group is required.

Intervention

A systematic review of the literature has been conducted in order to make sure that the telemedicine management is informed by evidence. Further, focus group interviews have been conducted both among patient groups and among health professionals, to ensure that the intervention is based on expert consensus.

The software used in the telemedicine intervention will be based on the established generic Patient Reported Outcome (PRO) system, WestChronic, which was developed in 2004 for collection of PRO data for research purposes in clinical epidemiological studies. WestChronic supports dynamic dual mode data collection with web or paper forms as well as communication to the patient with personalized postal letters, e-mails, and text messages. All information regarding implementations, items and questionnaires, communication, users, and patients resides in tables in a Structured Query Language (SQL) database, and all administration of implementations, questionnaires, users, and patients is supported by the server software and carried out in browser-windows. The software interphase serves a dual purpose: a) to be a customized communication tool between the patients and the health professionals, and b) to serve as decision support for the health professionals through the incorporation of a validated disease self-assessment tool.

Decision support, the Flare instrument

The Flare instrument (FI) serves as decision support for assessing disease activity in RA during the telemedicine intervention.

FI is a 12-item questionnaire where patients are asked to express their degree of agreement about different statements concerning disease activity on a 10-point likert scale. Six items concerns joint symptoms (tenderness, stiffness and pain) and six items is concerning general symptoms. When scoring FI it is possible to compute a FI total score (all 12 items) or a subscale for joint or general symptoms, respectively.

The instrument is translated into Danish according to the International Quality of Life Asessment (IQULA) method. It is validated in a cross sectional study among 100 consecutive patients from the outpatient clinic at Department of Rheumatology, Aarhus University Hospital, using DAS28 as the gold standard (unpublished data).

Execution

After randomization patients will be allocated to one of the three treatment arms: Telemedicine, doctor (TD), Telemedicine, Nurse (TN) or control in week 0, 13, 26, 39 and 52. The telemedicine consultation will be based on a telephone consultation. The consultation will follow a predefined consultation checklist.

Patients allocated to TD or TN, who has expressed a desire to complete questionnaires in webform, will receive a letter a week before the consultation to remind them that they must assess their disease activity through the software interphase, within the next couple of days. Patients, who have expressed a wish to fill in questionnaires in paper form, will receive the questionnaire a week before the consultation and asked to return it to WestChronic immediately after completion. A chasing procedure will be carried out in case of non-respondence. Two reminders will be send to the patients over a period of four weeks and continuous non-respondence will hereafter lead to exclusion from the study.

During telephone consultation, updated clinical test results will be available through the electronic medical system. Acute consultations will be performed and registered in all three groups as needed.

Statistics

Comparisons between groups will be made with the Fisher exact test for dichotomous responses and the Mann-Whitney U test for non-dichotomous responses. Changes over time will be analyzed with McNemar's test for dichotomous responses and Wilcoxon signed rank sum test for non-dichotomous responses. Data will be reported as a mean (SD) for variables in which normal distribution is found; otherwise data will be reported as the median ((interquartile range (IQR)).

Data will be analyzed using both "intention to treat" and per protocol. In case of missing data multiple imputations will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis according to the criteria's defined by the American College of Rheumatology, 1987, with a disease duration >= 2 years.

Exclusion Criteria:

* Patients unable to answer a questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score-CRP (DAS28, CRP) | One year
  RA disease activity is measured using DAS28, CRP. This score includes: tender and swollen joint count together with the patient's global assessment, report of physical functioning, the measurement of an acute-phase reactant. The DAS28 score run from 0-9.4 and RA disease activity is defined as followed: DAS28< 3.2: mild disease activity, DAS28 >3.2-< 5.1: moderate disease activity, DAS28 >5.1: high disease activity.

SECONDARY OUTCOMES:
Self-efficacy | One year
  Measured by the Generalized Self-Efficacy Scale (GSE), a 10-item scale with a score for each question ranging from 1 to 4. Higher scores indicate stronger patient's belief in self-efficacy.
  The GSE is designed to assess optimistic self-beliefs used to cope with a variety of demands in life. The scale was designed to assess self efficacy, i.e., the belief that one's actions are responsible for successful outcomes.
X Ray, hand and feet | one year
  Erosive changes

OTHER OUTCOMES:
The Flare Instrument (FI) | weeks 13, 26, 39 and 52
  A 12 item questionnaire where patients are asked to express their degree of agreement about different statements concerning disease activity on a 10-point likert scale. Six items concerns joint symptoms (tenderness, stiffness and pain) and six items is concerning general symptoms. When scoring FI it is possible to compute a FI total score (all 12 items) or a subscale for joint or general symptoms, respectively.
Quality of life (EQ5D) | one year
  EQ5D consists of a questionnaire and a VAS and is designed to measure well-being as well as illness
Health assessment Questionnaire | Weeks 13, 26, 39, 52
  Measures level of function among patients with arthritis

CONTACTS AND LOCATIONS:
Overall Officials: Annette de Thurah, MPH, Ph.D, Principal Investigator — Department of Rheumatology, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Rheumatology, Aarhus University Hospital, Aarhus
  - Department of Rheumatology, Silkeborg Regional Hospital, Silkeborg

REFERENCES:
- [Derived] de Thurah A, Stengaard-Pedersen K, Axelsen M, Fredberg U, Schougaard LMV, Hjollund NHI, Pfeiffer-Jensen M, Laurberg TB, Tarp U, Lomborg K, Maribo T. Tele-Health Followup Strategy for Tight Control of Disease Activity in Rheumatoid Arthritis: Results of a Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 Mar;70(3):353-360. doi: 10.1002/acr.23280. Epub 2018 Jan 23. PMID 28511288